CLINICAL TRIAL: NCT05665062
Title: A Phase 1 Study to Evaluate the Safety and Tolerability of a Combination Autologous CD19 CAR T Cell Therapy (SYNCAR-001 + STK-009) in Subjects With Relapsed or Refractory CD19+ Hematologic Malignancies
Brief Title: Autologous CD19 CAR-T Cell Therapy (SYNCAR-001) + Orthogonal IL-2 (STK-009) in Subjects With CD19+ Hematologic Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Synthekine (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STK-009-101
Record Dates: First submitted 2022-12-08; First posted 2022-12-27 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: CLL/SLL; NHL; Mantle Cell Lymphoma; Follicular Lymphoma; Large B-cell Lymphoma; Indolent B-Cell Non-Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma
Keywords: CART; CD19-CART; Chimeric antigen receptor; IL-2
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SYNCAR-001 + STK-009 Cohort A (Experimental): Dose escalation: A single fixed dose of autologous SYNCAR-001 CAR-T intravenously (IV) will be administered in combination with repeated sequential ascending doses of STK-009 subcutaneously (SC)
  Dose expansion: A single fixed dose of autologous SYNCAR-001 CAR-T IV will be administered in combination with repeated doses of STK-009 SC at the RP2D
  Interventions: Drug: SYNCAR-001; Drug: STK-009; Drug: Cyclophosphamide; Drug: Fludarabine
- SYNCAR-001 + STK-009 Cohort B (Experimental): Dose escalation: A single fixed dose of autologous SYNCAR-001 CAR-T intravenously (IV) will be administered in combination with repeated sequential ascending doses of STK-009 subcutaneously (SC)
  Dose expansion: A single fixed dose of autologous SYNCAR-001 CAR-T IV will be administered in combination with repeated doses of STK-009 SC at the RP2D
  Interventions: Drug: SYNCAR-001; Drug: STK-009

INTERVENTIONS:
Drug: SYNCAR-001 — SYNCAR-001 is an autologous CD19-targeted CAR-T with co-expression of hoRb
Drug: STK-009 — STK-009 is a human orthogonal IL-2 cytokine selective for SYNCAR-001 CAR-T cells expressing hoRb
Drug: Cyclophosphamide — lymphodepletion
  Arms: SYNCAR-001 + STK-009 Cohort A
Drug: Fludarabine — lymphodepletion
  Arms: SYNCAR-001 + STK-009 Cohort A

SUMMARY:
This is a first-in-human phase 1 study of SYNCAR-001 + STK-009 in patients with CD19+ hematologic malignancies.

DETAILED DESCRIPTION:
SYNCAR-001 + STK-009 is a 2-component human orthogonal (ho) IL-2 receptor-ligand cell therapy consisting of (1) SYNCAR-001, a CD19-directed chimeric antigen receptor T cell (CAR-T) co-expressing an engineered IL-2 beta receptor (hoRb); and (2) STK-009, an engineered pegylated IL-2 cytokine (hoIL-2) selective for hoRb. The study will follow a 3+3 design during dose escalation. Cohort A will enroll subjects to SYNCAR-001 + STK-009 with lymphodepletion. At Dose Level 3, a separate dose escalation cohort will be introduced to enroll subjects to SYNCAR-001 + STK-009 without lymphodepletion (Cohort B). Subsequent dose expansions will enroll subjects at the RP2D for each cohort.

ELIGIBILITY:
Selected Inclusion Criteria:

1. Histologically confirmed relapsed/refractory hematologic malignancies, including Chronic Lymphocytic Lymphoma (CLL/SLL) and selected Non-Hodgkin's Lymphoma (NHL)
2. Prior or current documentation of CD19 expression or high likelihood of CD19 expression based on disease histology
3. No signs of symptoms of central nervous system (CNS) disease or detectable evidence of CNS or meningeal disease on magnetic resonance imaging (MRI) at the time of screening

Selected Exclusion Criteria:

1. Prior CD19 directed therapy including CD19 CARTs
2. Prior allogeneic hematopoietic stem cell transplant within 6 months of enrollment
3. Prior autologous hematopoietic stem cell transplant within 6 weeks of enrollment.
4. Presence of GVHD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04-23 (Actual); Primary Completion 2026-06-24 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) | Up to 28 days post infusion (SYNCAR-001+STK-009)
  Incidence of adverse events (AEs) meeting protocol defined DLT criteria and determination of the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of STK-009 in combination with a fixed dose of SYNCAR-001
Adverse events | Up to 24 months post infusion (SYNCAR-001+STK-009)
  Assess the safety and tolerability of STK-009 in combination with SYNCAR-001 by review of AEs

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 24 months post infusion (SYNCAR-001+STK-009)
  The ORR to treatment with SYNCAR-001 + STK-009
Duration of Response (DOR) | Up to 24 months post infusion (SYNCAR-001+STK-009)
  To evaluate the duration of anti-cancer response after SYNCAR-001 + STK-009 administration.
Progression Free Survival (PFS) | Up to 24 months post infusion (SYNCAR-001+STK-009)
  The time from the SYNCAR-001 administration date to the date of disease progression per Lugano Classification or iwCLL or death from any cause, whichever occurs earlier.
Area under the curve (AUC) | Up to 24 months post infusion (SYNCAR-001+STK-009)
  The quantification of the cumulative amount of drug over time.
Maximum Concentration (Cmax) | Up to 24 months post infusion (SYNCAR-001+STK-009)
  To identify the maximum (peak) drug concentration dosing.
Time of maximum concentration | Up to 24 months post infusion (SYNCAR-001+STK-009)
  The time to reach maximum (peak) drug concentration after dosing.
Immunogenicity | Up to 24 months post infusion (SYNCAR-001+STK-009)
  Immunogenicity will be assessed by summarizing the number of patients who develop detectable anti-STK-009 and/or anti-SYNCAR-001 anti-drug antibodies (ADAs)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - City of Hope, Duarte, California
  - Roswell Park, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No